CLINICAL TRIAL: NCT01837095
Title: A Phase I Dose Escalation Study of POL6326 With Eribulin in Patients With Relapsed, Triple Negative and Hormone Refractory ER Positive Metastatic Breast Cancer
Brief Title: Dose Escalation of POL6326 in Combination With Eribulin in Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Polyphor Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POL-7
Record Dates: First submitted 2013-04-02; First posted 2013-04-22 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Metastatic Breast Cancer
Keywords: Overall survival; Progression free survival
MeSH Terms: conditions — Breast Neoplasms | interventions — balixafortide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- POL6326 (Experimental): POL6326 will be given by i.v. infusion over 2 hours. Treatment will occur on days prior to, on the day of and on days after treatment with eribulin
  Interventions: Drug: POL6326

INTERVENTIONS:
Drug: POL6326 — POL6326 will be given by i.v. infusion over 2 hours. Treatment will occur on days prior to, on the day of and on days after treatment with eribulin

SUMMARY:
POL6326 will be given by i.v. infusion over 2 hours. Treatment will occur on days prior to, on the day of and on days after treatment with eribulin. Different doses and dosing frequencies will be investigated

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive cancer of the breast.
* Presence of at least one measurable lesion per RECIST 1.1 criteria
* Stage IV disease by AJCC criteria (7th edition).
* HER2 negative (IHC 0,1 or FISH HER2:CEP17 ratio < 2.0)
* Must have had treatment with at least 2 but no more than 3 previous regimens in the metastatic setting. Previous treatment must have included an anthracycline and taxane in either the adjuvant or metastatic setting.
* At least 21 days from the completion of any previous cytotoxic chemotherapy or biological therapy at time of initiation of POL6326.
* ECOG performance status < 2

Exclusion Criteria:

* Previously received eribulin.
* Peripheral neuropathy > Grade 2.
* Receipt of any other investigational agent within the 28 days prior to Day 1.
* Receipt of colony stimulating factor filgrastim, pegfilgrastim, or sargramostim within 14 days prior to Day 1.
* Radiation therapy within the 14 days prior to Day 1.
* Severe concurrent illness or psychiatric illness/social situation that would limit compliance with study requirements.
* History of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Pregnant or breastfeeding.
* Known HIV positivity on combination antiretroviral therapy; these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2013-06; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of POL6326 in combination with eribulin in patients with metastatic breast cancer | 6 months
  Incidence and severity of adverse events and serious adverse events of the combination of POL6326 and eribulin when compared to the adverse event profile of eribulin alone

SECONDARY OUTCOMES:
Response rate of treatment with POL6326 and eribulin in patients with metastatic breast cancer | 12-24 months
  Determination of the complete response (CR) and partial response (PR) in patients treated with the combination of POL6326 and eribulin

CONTACTS AND LOCATIONS:
Locations (12):
- United States (5):
  - St Luke's Cancer Institute, Kansas City, Kansas
  - Washington University School of Medicine, Division of Oncology, St Louis, Missouri
  - 'Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Weill Cornell Breast Center, New York, New York
  - Vanderbilt University School of Medicine, Nashville, Tennessee
- Spain (7):
  - Hospital del Mar, Barcelona
  - Hospital Quiron Barcelona, Barcelona
  - Hospital Vall d'Hebrón, Barcelona
  - Instituto Catalàn de Oncologia L'Hospitalet, L'Hospitalet de Llobregat
  - HGUG Marañón, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Cinico Universitario de ValenciaValencia, Valencia

REFERENCES:
- [Derived] Pernas S, Martin M, Kaufman PA, Gil-Martin M, Gomez Pardo P, Lopez-Tarruella S, Manso L, Ciruelos E, Perez-Fidalgo JA, Hernando C, Ademuyiwa FO, Weilbaecher K, Mayer I, Pluard TJ, Martinez Garcia M, Vahdat L, Perez-Garcia J, Wach A, Barker D, Fung S, Romagnoli B, Cortes J. Balixafortide plus eribulin in HER2-negative metastatic breast cancer: a phase 1, single-arm, dose-escalation trial. Lancet Oncol. 2018 Jun;19(6):812-824. doi: 10.1016/S1470-2045(18)30147-5. Epub 2018 Apr 26. PMID 29706375